CLINICAL TRIAL: NCT04841616
Title: Multicentered Prospective Randomized Controlled Trial On Contrast-Enhanced Harmonic Endoscopic Ultrasound (CH_EUS) Vs Conventional EUS-Guided Fine Needle Biopsy (FNB) For Solid Pancreatic Lesions
Brief Title: Multicentered Prospective Randomized Controlled Trial For Solid Pancreatic Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Charing Chong, MD, Dr, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CREC2020.496
Record Dates: First submitted 2021-03-30; First posted 2021-04-12 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Pancreas Neoplasm
Keywords: Contrast-Enhanced EUS; FNB; Solid Pancreatic Lesions
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contrast-enhanced EUS (CH-EUS) Arm (Experimental): After initial evaluation, 2.5ml of second-generation contrast media, SonoVue (Bracco, Ceriano Laghetto, Italy), will be injected. After infusion, the point of puncture will be determined when the parenchyma of the pancreas was enhanced. The contrast-enhanced area was identified and then the biopsy was directed toward that area, while avoiding unenhanced (i.e. necrotic) areas and not changing the target lesion. Rest of the procedure is identical with that in conventional EUS arm.
  Interventions: Procedure: Contrast-Enhanced Harmonic Endoscopic Ultrasound
- Conventional EUS Arm (Active Comparator): Patients will undergo EUS FNB with the 22-gauge FNB needle (Acquire®, Boston Scientific Natick, MA). After each pass, the needle is removed and the stylet will be introduced into the needle to extrude any aspirated material on a glass slide for inspection of the presence of a macroscopic visible core (MVC). The total length of the MVC will be measured before placement into a formalin bottle. EUS-FNB is completed if the obtained MVC is longer than 4mm and deemed adequate by endoscopist. If the obtained MVC is < 4mm, the procedure is repeated until a MVC of ≥ 4mm is obtained and deemed adequate by endoscopist. A maximum of 7 passes is allowed
  Interventions: Procedure: Endoscopic Ultrasound -Guided Fine Needle Biopsy

INTERVENTIONS:
Procedure: Endoscopic Ultrasound -Guided Fine Needle Biopsy — Patients will undergo EUS FNB with the 22-gauge FNB needle (Acquire®, Boston Scientific Natick, MA). After each pass, the needle is removed and the stylet will be introduced into the needle to extrude any aspirated material on a glass slide for inspection of the presence of a macroscopic visible core (MVC). The total length of the MVC will be measured before placement into a formalin bottle. EUS-FNB is completed if the obtained MVC is longer than 4mm and deemed adequate by endoscopist. If the obtained MVC is < 4mm, the procedure is repeated until a MVC of ≥ 4mm is obtained and deemed adequate by endoscopist. A maximum of 7 passes is allowed.
  Arms: Conventional EUS Arm
Procedure: Contrast-Enhanced Harmonic Endoscopic Ultrasound — After initial evaluation, 2.5ml of second-generation contrast media, SonoVueTM (Bracco, Ceriano Laghetto, Italy), will be injected. After infusion, the point of puncture will be determined when the parenchyma of the pancreas was enhanced. The contrast-enhanced area was identified and then the biopsy was directed toward that area, while avoiding unenhanced (i.e. necrotic) areas and not changing the target lesion. Rest of the procedure is identical with that in conventional EUS arm.
  Arms: Contrast-enhanced EUS (CH-EUS) Arm

SUMMARY:
Endoscopic ultrasound (EUS) is an indispensable tool for tissue acquisition for pancreatic lesions. Fine needle aspiration (FNA) is once considered as the first line diagnostic method especially when rapid on-site evaluation (ROSE) by cytopathologist is available.

However, FNA alone has several limitations including inadequate acquisition of cells, and unable to provide core tissue for further histological analysis. Furthermore, ROSE is not available in many endoscopic centres due to limited resources. Endosonographers around the world, are discovering methods to overcome the limitations, including the use of new on-site evaluation technique by endoscopists, new fine-needle biopsy (FNB) needles, contrast-enhanced harmonic EUS-guided FNB.

In this study, the investigators propose to compare the diagnostic performance between contrast-enhanced EUS-guided FNB versus conventional EUS-guided FNB technique with an aim to define the best EUS-guided tissue acquisition technique in the absence of ROSE. Results obtained from this research is expected to have significant impact in providing new insights on the best EUS-guided tissue acquisition method. It may replace FNA with ROSE as the gold standard for EUS-guided tissue acquisition in an affordable manner. It will also save the patients from unnecessary procedures and fasten the treatment pathways.

DETAILED DESCRIPTION:
Seicean et al, in a prospective study, evaluated the diagnostic accuracy of EUS-FNA with CH-EUS using SonoVueTM versus EUS-FNA without CH-EUS. They found that the diagnostic accuracy of EUS-FNA with CH-EUS was higher than that of EUSFNA without CH-EUS (86.5% vs 78.4%). However, the difference did not reach the threshold required for statistical significance. Also, only FNA, but not FNB, was performed in this study.

The FNB needle was introduced to further improve upon EUS guided tissue sampling. It is designed to collect a larger amount of core sample tissue with preserved histological architecture for further analysis, including molecular analysis. Also the FNB needle has been shown to obtain samples with higher cellularity compared to the standard FNA needles. Compared with EUS-FNA, EUS-FNB had a better specimen adequacy, higher diagnostic accuracy, and fewer number of needle passes but no increase in complications rate.

The technique of macroscopic on-site evaluation (MOSE) has recently been advocated for estimating the adequacy of a core specimen obtained by EUS for histological diagnosis. MOSE involves immediate examination of the FNB specimen for the presence of a "macroscopic visible core" (MVC), which is defined as whitish or yellowish pieces of tissue with an apparent bulk. The total length of the MVC is then measured and the optimal cut-off MVC length was 4 mm. This study demonstrated that EUS-FNB with MOSE provided comparable diagnostic yield as EUS-FNB without MOSE (92.6% vs 89.3%) with fewer numbers of passes.

Puncturing avascular or necrotic area of a tumour could be the major reason of false negative rate during EUS-guided FNB. Contrast-enhanced harmonic EUS (CH-EUS) can define avascular or necrotic area inside a tumour which may improve the false negative rate during EUS-FNB. In this study, the investigators aim to evaluate the diagnostic performance of CH-EUS-guided FNB with MOSE for solid pancreatic masses. The investigators expect the study will define the best EUS-guided tissue acquisition technique in the absence of ROSE and replace FNA with ROSE as gold standard for tissue sampling for solid pancreatic masses.

ELIGIBILITY:
Inclusion Criteria:

* referred for EUS-guided tissue acquisition for solid pancreatic lesions greater than 1cm in the largest diameter.

Exclusion Criteria:

* with coagulopathy, altered anatomy, contraindications for conscious sedation, pregnancy
* who cannot provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
False negative rate | up to 6 months

SECONDARY OUTCOMES:
sensitivity | up to 6 months
specificity | up to 6 months
procedural time | within 1 day
  minute
procedure-related complications | up to 6 months
  Bleeding, perforation, etc
the need to repeat procedure | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ching Ning Chong, Principal Investigator — CUHK
Locations (1):
- Department of Surgery; The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Strand DS, Jeffus SK, Sauer BG, Wang AY, Stelow EB, Shami VM. EUS-guided 22-gauge fine-needle aspiration versus core biopsy needle in the evaluation of solid pancreatic neoplasms. Diagn Cytopathol. 2014 Sep;42(9):751-8. doi: 10.1002/dc.23116. Epub 2014 Feb 18. PMID 24550162
- [Background] Aadam AA, Wani S, Amick A, Shah JN, Bhat YM, Hamerski CM, Klapman JB, Muthusamy VR, Watson RR, Rademaker AW, Keswani RN, Keefer L, Das A, Komanduri S. A randomized controlled cross-over trial and cost analysis comparing endoscopic ultrasound fine needle aspiration and fine needle biopsy. Endosc Int Open. 2016 May;4(5):E497-505. doi: 10.1055/s-0042-106958. PMID 27227104
- [Background] Lee YN, Moon JH, Kim HK, Choi HJ, Choi MH, Kim DC, Lee TH, Cha SW, Cho YD, Park SH. Core biopsy needle versus standard aspiration needle for endoscopic ultrasound-guided sampling of solid pancreatic masses: a randomized parallel-group study. Endoscopy. 2014 Dec;46(12):1056-62. doi: 10.1055/s-0034-1377558. Epub 2014 Aug 6. PMID 25098611
- [Background] Iwashita T, Yasuda I, Mukai T, Doi S, Nakashima M, Uemura S, Mabuchi M, Shimizu M, Hatano Y, Hara A, Moriwaki H. Macroscopic on-site quality evaluation of biopsy specimens to improve the diagnostic accuracy during EUS-guided FNA using a 19-gauge needle for solid lesions: a single-center prospective pilot study (MOSE study). Gastrointest Endosc. 2015 Jan;81(1):177-85. doi: 10.1016/j.gie.2014.08.040. Epub 2014 Oct 29. PMID 25440688
- [Background] Seicean A, Badea R, Moldovan-Pop A, Vultur S, Botan EC, Zaharie T, Saftoiu A, Mocan T, Iancu C, Graur F, Sparchez Z, Seicean R. Harmonic Contrast-Enhanced Endoscopic Ultrasonography for the Guidance of Fine-Needle Aspiration in Solid Pancreatic Masses. Ultraschall Med. 2017 Apr;38(2):174-182. doi: 10.1055/s-0035-1553496. Epub 2015 Aug 14. PMID 26274382
- [Background] Fuccio L, Larghi A. Endoscopic ultrasound-guided fine needle aspiration: How to obtain a core biopsy? Endosc Ultrasound. 2014 Apr;3(2):71-81. doi: 10.4103/2303-9027.123011. PMID 24955336
- [Background] Iglesias-Garcia J, Poley JW, Larghi A, Giovannini M, Petrone MC, Abdulkader I, Monges G, Costamagna G, Arcidiacono P, Biermann K, Rindi G, Bories E, Dogloni C, Bruno M, Dominguez-Munoz JE. Feasibility and yield of a new EUS histology needle: results from a multicenter, pooled, cohort study. Gastrointest Endosc. 2011 Jun;73(6):1189-96. doi: 10.1016/j.gie.2011.01.053. Epub 2011 Mar 21. PMID 21420083
- [Background] Yang MJ, Yim H, Hwang JC, Lee D, Kim YB, Lim SG, Kim SS, Kang JK, Yoo BM, Kim JH. Endoscopic ultrasound-guided sampling of solid pancreatic masses: 22-gauge aspiration versus 25-gauge biopsy needles. BMC Gastroenterol. 2015 Sep 29;15:122. doi: 10.1186/s12876-015-0352-9. PMID 26419845
- [Background] Kin T, Katanuma A, Yane K, Takahashi K, Osanai M, Takaki R, Matsumoto K, Gon K, Matsumori T, Tomonari A, Maguchi H, Shinohara T, Nojima M. Diagnostic ability of EUS-FNA for pancreatic solid lesions with conventional 22-gauge needle using the slow pull technique: a prospective study. Scand J Gastroenterol. 2015 Jul;50(7):900-7. doi: 10.3109/00365521.2014.983155. Epub 2015 Mar 2. PMID 25732902
- [Background] Teoh AYB, Serna C, Penas I, Chong CCN, Perez-Miranda M, Ng EKW, Lau JYW. Endoscopic ultrasound-guided gallbladder drainage reduces adverse events compared with percutaneous cholecystostomy in patients who are unfit for cholecystectomy. Endoscopy. 2017 Feb;49(2):130-138. doi: 10.1055/s-0042-119036. Epub 2016 Nov 22. PMID 27875855
- [Background] Teoh AY, Ng EK, Chan SM, Lai M, Moran S, Binmoeller KF, Moon JH, Ho KY. Ex vivo comparison of the lumen-apposing properties of EUS-specific stents (with video). Gastrointest Endosc. 2016 Jul;84(1):62-8. doi: 10.1016/j.gie.2015.11.041. Epub 2015 Dec 10. PMID 26684601
- [Background] Teoh AYB, Chong CCN, Leung WW, Chan SKC, Tse YK, Ng EKW, Lai PBS, Wu JCY, Lau JYW. Electroacupuncture-reduced sedative and analgesic requirements for diagnostic EUS: a prospective, randomized, double-blinded, sham-controlled study. Gastrointest Endosc. 2018 Feb;87(2):476-485. doi: 10.1016/j.gie.2017.07.029. Epub 2017 Jul 24. PMID 28750840
- [Background] Chong CCN, Tang RSY, Wong JCT, Chan AWH, Teoh AYB. Endoscopic ultrasound of pancreatic lesions. J Vis Surg. 2016 Jul 22;2:119. doi: 10.21037/jovs.2016.07.10. eCollection 2016. PMID 29399505
- [Background] Teoh AY, Chong CC, Chan AW, Lau JY. EUS-guided alcohol injection of pancreatic neuroendocrine tumor. Gastrointest Endosc. 2015 Jul;82(1):167. doi: 10.1016/j.gie.2015.01.047. Epub 2015 Apr 22. No abstract available. PMID 25910658
- [Background] Chong CCN, Teoh AYB, Tang RSY, Chan AWH, Ng EKW, Lai PBS. EUS-FNA using 22G nitinol or ProCore needles without on-site cytopathology. Endosc Ultrasound. 2018 Jan-Feb;7(1):56-60. doi: 10.4103/eus.eus_113_17. PMID 29451170